CLINICAL TRIAL: NCT03996226
Title: A Phase 1 Food-Effect Study of E7386 in Healthy Subjects
Brief Title: A Food-Effect Study of E7386 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: E7386-A001-001
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-06

CONDITIONS: Food Effect in Healthy Participants
Keywords: Healthy Participants; E7386; Bioavailability; Food Effect
MeSH Terms: interventions — E-7386

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E7386: Fed + Fast (Experimental): Participants will receive a single oral dose of E7386 tablet in fed condition on Day 1 of treatment period 1 followed by a single oral dose of E7386 tablet in fasted condition on Day 8 of treatment period 2. A washout period of 7 days will be maintained between the 2 treatment periods.
  Interventions: Drug: E7386
- E7386: Fast + Fed (Experimental): Participants will receive a single oral dose of E7386 tablet in fasted condition on Day 1 of treatment period 1 followed by a single oral dose of E7386 tablet in fed condition on Day 8 of treatment period 2. A washout period of 7 days will be maintained between the 2 treatment periods.
  Interventions: Drug: E7386

INTERVENTIONS:
Drug: E7386 — E7386 oral tablets.

SUMMARY:
The primary objective of this study is to determine the effect of food in healthy participants on the bioavailability of E7386 following single dose administration with and without a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, healthy participants at the time of informed consent.
2. Body Mass Index (BMI) greater than (>) 18 and less than or equal to (<=) 30 kilogram per square meter (kg/m^2) at Screening.

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 international units per litre (IU/L) or equivalent units of ß-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
2. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

     1. total abstinence (if it is their preferred and usual lifestyle)
     2. an intrauterine device or intrauterine hormone-releasing system
     3. a contraceptive implant
     4. an oral contraceptive (with additional barrier method) (Participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation)
     5. have a vasectomized partner with confirmed azoospermia
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
3. Males who have not had a successful vasectomy (confirmed azoospermia) and their female partners meet the exclusion criteria No: 2, above. If the female partner is pregnant, then males who do not agree to use Barrier contraception (latex or synthetic condoms) throughout the study period and for 90 days after study drug discontinuation. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
5. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
6. Any history of major surgery, e.g., intestinal resections, hepatectomy, nephrectomy, digestive organ resection that may affect absorption, metabolism or excretion of E7386.
7. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, electrocardiogram (ECG) finding, or laboratory test results that require medical treatment at Screening
8. Clinically significant ECG abnormality including a marked baseline prolongation of QT/corrected QT interval (QTc) (example: repeated demonstration of a QTc interval greater than (>) 500 milliseconds [msec]), or a family history of prolonged QTc syndrome or sudden death
9. History of drug or alcohol misuse within 6 months prior to Screening, or who had a positive urine drug test at Screening or Baseline
10. Diagnosed with acquired immune deficiency syndrome, or test positive for human immunodeficiency virus (HIV) at screening
11. Active viral hepatitis (A, B or C) as demonstrated by positive serology at Screening
12. Use of prescription drugs within 4 weeks prior to dosing
13. Intake of over-the-counter medications within 2 weeks prior to dosing
14. Intake of caffeinated beverages or food within 72 hours prior to dosing
15. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing
16. Participated in another clinical trial less than 4 weeks prior to dosing or was currently enrolled in another clinical trial
17. Consumed grapefruit, starfruit, Seville oranges or their products within 7 days prior to dosing
18. Consumed herbal preparations/medications including but not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng within 7 days prior to dosing
19. Allergic to E7386 or any of the tablet's ingredients
20. Known history of clinically significant drug or food allergies, or presently experiencing significant seasonal or perennial allergy at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for E7386 | Day 1: 0-48 hours; Day 8: 0-48 hours
Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for E7386 | Day 1: 0-48 hours; Day 8: 0-48 hours
AUC0-t: AUC 0-t: Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration for E7386 | Day 1: 0-48 hours; Day 8: 0-48 hours
AUC0-inf: Area Under the Plasma Concentration-time Curve from Time 0 to Infinite Time for E7386 | Day 1: 0-48 hours; Day 8: 0-48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.